CLINICAL TRIAL: NCT04794959
Title: Detection of Bowel Hypoperfusion Among Chronic Mesenteric Ischemia Patients During Meal Digestion Using Dual-Energy CT (DECT) - A Pilot Study.
Brief Title: A Pilot Study on the Using a Newer Computed Tomography (CT) Based Technique for the Detection of Altered Bowel Blood Flow Among Patients Suffering From Chronic Mesenteric Ischemia During Meal Digestion.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jack Xu, MD, PhD-student, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-20066374
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Bowel; Ischemic, Chronic; Tomography, X-Ray Computed; Dual-energy CT
MeSH Terms: conditions — Ischemia; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Dual-energy CT — CMI patients planned for endovascular stent placement will be contacted and informed about this study prior to their procedure. If they wish to take part in the study, then a date for a pre-operative DECT scan will be arranged. Before scanning the patient will be given a standardized calorie dense drink (Nutridrink). This will take place one week prior to their surgical procedure. Following the surgical procedure, the patient will undergo another DECT scan before discharge.

SUMMARY:
Chronic meseteric ischemia (CMI) is a disease characterized by an insufficient blood supply to the intestines due to a narrowing (stenosis) of one or multiple intestinal arteries. The primary symptom is abdominal pain especially during meal digestion. Currently the diagnosis of CMI is heavily reliant on the exclusion of differential diagnoses. With this study we wish to evaluate whether a newer CT technology called dual-energy CT (DECT) may be able to visualize this altered blood flow during meal consumption.

DETAILED DESCRIPTION:
CMI is a relatively rare condition mainly affecting elderly patients >60 years old. CMI is characterized by an insufficient blood supply to the intestines due to a narrowing (stenosis) of one or multiple intestinal arteries. The main symptoms associated with CMI are abdominal pain following mealtimes and weight loss. Diagnosis for CMI is difficult as >10% of all elderly patients have stenotic changes in their intestinal arteries, however only a fraction of these patients are symptomatic. The diagnosis of CMI is therefore mainly based on the clinical history and evaluation. The challenging diagnosis is most likely the main contributing factor to why five to 19% of patients experience no symptomatic relief following surgical treatment. The surgical treatment consists of either open surgical bypass or, more commonly, endovascular stent placement, opening the stenotic artery.

Endovascular stent placement for patients with symptomatic CMI is a common procedure at the Department of Diagnostic Radiology and Department of Vascular Surgery, Rigshospitalet, with approximately 60 patients undergoing the procedure annually. Patients undergo a preoperative CT scan including a non-contrast and arterial phase scan to evaluate the abdominal arterial vessels and the degree of stenosis, however the bowel wall is not routinely evaluated. This is mainly due to the fact that mesenteric blood flow is adequate during times of fasting, however insufficient blood flow may occur at times of peak demand i.e. during digestion of a meal.

DECT has shown improved conspicuity for bowel ischemia using monoenergetic images and allows for iodine selective maps which have been used in the evaluation of pulmonary emboli.

To our knowledge, there are no current studies that have investigated applications of DECT in the evaluation of CMI. We intend to investigate whether it is possible to visualize bowel hypoperfusion using DECT following administration of a standardized meal.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed CMI patients planned for endovascular stent placement treatment

Exclusion Criteria:

* Noncomplete dataset
* Allergies to contrast agents
* Suboptimal CT images
* Issues related to the administration of the calorie drink

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Pre- and post-operative DECT scans on CMI patients | 10 days

IPD SHARING:
Plan to Share IPD: No